CLINICAL TRIAL: NCT00619996
Title: Phase II Study of Sorafenib (Bay 43-9006) and Docetaxel in Metastatic Prostate Cancer
Brief Title: Study of Sorafenib and Docetaxel in Metastatic Prostate Cancer
Acronym: P1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Italian Trial in Medical Oncology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PISAUNO
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Last update posted 2009-02-26 (Estimated); Status verified 2009-02

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Sorafenib; Nexavar; Docetaxel; Pisa; Ricci
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Sorafenib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Sorafenib (Nexavar); Drug: Docetaxel

INTERVENTIONS:
Drug: Sorafenib (Nexavar) — Sorafenib 400 mg bid orally continuously
  Sorafenib will be administered from the start of treatment in combination with Docetaxel until progression of disease.
  Other Names: TRATTAMENTO
Drug: Docetaxel — Docetaxel 75 mg/mq ev g1 every 21 days. Docetaxel will be administered for a maximum of 9 cycles.

SUMMARY:
The purpose of this study is to use Sorafenib plus Docetaxel to evaluate pharmacodynamics (PD) in Patients with prostate cancer.

DETAILED DESCRIPTION:
Background Prostate cancer is the most common malignancy in men and the second leading cause of cancer death among males in the Western World. When tumors become refractory to androgen withdrawal therapy, chemotherapy represent a palliative treatment with an improvement on quality of life, particularly the combination of mitoxantrone and prednisone . This observation has led to numerous studies evaluating the potential use of new chemotherapeutic agents as Docetaxel in patients with metastatic androgen independent prostate cancer. Recently Docetaxel based regimens have shown an improvement in survival when compared with mitoxantrone in a phase III trial .

However the prognosis of these patients remains very poor and new effective tolerated approaches are needed to improve the results of chemotherapy.

Rationale In a recent study a Raf kinase inhibitor protein (RKIP) encoded by a suppressor gene was found to be responsible of the metastatic process; in fact the decreased RKIP expression was associated with increased invasive capability of prostate cancer cells, presumably though the activation of MEK and ERK by phosphorilation .

Sorafenib, a novel signal transduction inhibitor, prevents tumor cell proliferation and angiogenesis blocking Raf/Mek/Erk pathway at the level of Raf kinase and tyrosine kinase receptors VEGFR-2 and PDGFR.

In a phase I study the combination of docetaxel and Sorafenib was evaluated in prostate and other tumors . The treatment was well tolerated and one partial response (4%) and 12 stable disease (50%) were reported.

According to these data we designed a phase II study to evaluate the association of Sorafenib and Docetaxel in metastatic prostate cancer

Simon's Optimal two-stage design for phase II clinical trial will be applied to calculate the sample size that minimizes the expected number of patients to be accrued. The sample size will be calculated on the following assumptions: alpha error =0.05, beta error =0.20; PD (clinically uninteresting true no progressive disease rate) and P1 (sufficiently promising true no progressive disease rate) will be set at 60% and 80%. 11 patients will be enrolled in the first stage: if no progressive diseases are < 7 the accrual will be stopped and the drug's combination rejected. In the case of >= 7 no progressive diseases 32 more patients will be accrued at the second stage. The treatment will be accepted if >= 30 no progressive diseases out of 43 patients will be observed

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic hormone refractory prostate cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2007-03; Primary Completion 2008-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
N° of no progressive disease | 1 year

SECONDARY OUTCOMES:
ORR,Duration of responses,TTP,OS,PSA doubling time, PK-PD,of Sorafenib plus docetaxel,Baseline pERK concentration, phospho VEGF-R2 concentration, plasma proteomics and gene expression profiling on blood cells and tumor biopsy. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Dipartimento di Oncologia, dei Trapianti e delle Nuove Tecnologie in Medicina ... Indirizzo: via Roma, 55 - 56100 Pisa Tel. 050-2218690 - Fax. 050-2218685, Pisa, Pisa, Italy